CLINICAL TRIAL: NCT02190136
Title: Yoga Improves Aerobic Fitness, Glycemia and Mood State and Reduces Abdominal Obesity in Overweight Women: The PRISE Study
Brief Title: Yoga Improves Aerobic Fitness, Glycemia and Mood State and Reduces Abdominal Obesity
Acronym: PRISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Principal Investigator, Paul Arciero, Professor, Health and Exercise Sciences Department, Skidmore College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Yoga-0610-52
Record Dates: First submitted 2014-07-07; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Obesity; Insulin Resistance
Keywords: obesity; protein-rich whole foods diet; aerobic fitness; resistance training; stretching/yoga training; glycemia; mood state
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein whole foods (Active Comparator): Ingestion of 20-25 grams per serving consumed 4-6 times per day; 1 within an hour of waking in the morning and the other 2.5-3 hours apart during the day.
  Interventions: Other: Protein whole foods; Other: Protein Resistance Exercise Training; Other: Protein Stretching/Yoga Training
- Protein Resistance Exercise Training (Experimental): Ingestion of 4-6 protein-rich meals per day and 3 times per week of resistance functional training.
  Interventions: Other: Protein whole foods; Other: Protein Resistance Exercise Training
- Protein Stretching/Yoga Training (Experimental): Ingestion of Protein-rich diet 4-6 meals/day and stretching/yoga training 3 times per week
  Interventions: Other: Protein whole foods; Other: Protein Stretching/Yoga Training

INTERVENTIONS:
Other: Protein whole foods — Protein-rich whole foods consumed at 20-30 grams of protein at each of 4-6 meals per day
Other: Protein Resistance Exercise Training — Protein rich whole foods diet and resistance training 3 times per week for 11 weeks
  Arms: Protein Resistance Exercise Training; Protein whole foods
Other: Protein Stretching/Yoga Training — Protein-rich whole foods diet of 20-30 grams of protein at each of 4-6 meals per day with stretching/yoga training 3 times per week for 11 weeks
  Arms: Protein Stretching/Yoga Training; Protein whole foods

SUMMARY:
Stretching and flexibility exercise such as yoga and functional resistance exercise are two forms of exercise that are growing in popularity. However, they have not been scientifically tested to demonstrate their ability to improve body composition, fitness, heart and metabolic health, and mood state in overweight/obese women. The investigators hypothesize that during an 11 week intervention, both forms of exercise will improve body composition, heart and metabolic health and mood state.

DETAILED DESCRIPTION:
This study was a 11 week protein-rich whole food diet and exercise training intervention in middle aged overweight/obese women. Subjects were randomized into 3 groups: Protein-rich whole food only consumed as 20-25 grams per serving 4-6 per day (P); protein and resistance exercise training (R); and protein and stretching/yoga exercise training (S). All outcomes, including the primary outcomes of body composition and cardiometabolic biomarkers were measured at baseline (week 0) and post-intervention (week 12) in all study subjects.

ELIGIBILITY:
Inclusion Criteria:

* obese or overweight women
* between ages 25-60 and
* otherwise healthy

Exclusion Criteria:

* smokers,
* habitual exercisers

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Total and Regional Body Composition | baseline and 11 weeks
  Total and regional body composition was assessed by dual energy xray absorptiometry (DXA) at baseline and 11 weeks in all subjects

SECONDARY OUTCOMES:
Aerobic Fitness | baseline and 11 weeks
  VO2 max was assessed in each subject at baseline and 11 weeks

OTHER OUTCOMES:
Plasma Biomarkers | baseline and 11 weeks
  Insulin, glucose, and leptin was assessed in each subject at baseline and 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, PhD, Principal Investigator — Skidmore College
Locations (1):
- Human Nutrition and Metabolism Laboratory, Saratoga Springs, New York, United States

REFERENCES:
- [Derived] Ruby M, Repka CP, Arciero PJ. Comparison of Protein-Pacing Alone or With Yoga/Stretching and Resistance Training on Glycemia, Total and Regional Body Composition, and Aerobic Fitness in Overweight Women. J Phys Act Health. 2016 Jul;13(7):754-64. doi: 10.1123/jpah.2015-0493. Epub 2016 Feb 19. PMID 26901102